CLINICAL TRIAL: NCT04487132
Title: Impact of School Based Intervention on Motivation Towards Physical Activity and Psychosocial Outcomes Among Adolescents: A Randomized Control Trial
Brief Title: Impact of School Based Intervention on Motivation Towards Physical Activity and Psychosocial Outcomes Among Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Anmol Ayaz, principle investigator, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FJWU/Reg/2020
Record Dates: First submitted 2020-07-10; First posted 2020-07-27 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: School Based Intervention

STUDY DESIGN:
Intervention Model Description: Randomized control trial design will be used in this study to examine the impact of school-based intervention on motivation towards physical activity and psychosocial outcomes among adolescents. In trials with randomized and controlled design the effects of the study (school based intervention and psychosocial outcomes) are compared with those of a control group and the participants are randomly assigned to the two groups. In this interventional model Active physical education lessons and physical education plan will be carried out which includes, Physical activities 10 -15 minutes daily or at least 5 days in a week during the school timings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active physical education lessons and physical education plan (Active Comparator): Active physical education lessons and physical education plan provided to the controlled group
  Interventions: Behavioral: Active physical education lessons and physical education plan
- Recess or lunch time activities (Active Comparator): Preparing the playground by offering adequate spaces and games provided to the experimental group
  Interventions: Behavioral: Active physical education lessons and physical education plan; Behavioral: Recess or lunch time activities

INTERVENTIONS:
Behavioral: Active physical education lessons and physical education plan — Active physical education lessons and physical education plan Including importance of physical activity and health, and physical education plan; through lecture in classroom will be provided to the contyrolled group.
  Other Names: physical education plan
Behavioral: Recess or lunch time activities — group intervention will be provided ti the experimental group which includes Preparing the playground by offering adequate spaces and games.Developing games and teaching children to play in recess time at-least 10-15 minutes daily(i.e.sport games, traditional games) Placing a sheet in the classroom with some reminders about being active in recess time (i.e. using a poster board encouraging playing one of the selected games )
  Other Names: physical activities group intervention
  Arms: Recess or lunch time activities

SUMMARY:
This study examines the effect of self designed school-based interventions on physical activity and psychological outcomes (i.e., internalizing and externalizing behavioral symptoms, self-concept, and academic achievement among a community sample of adolescents from Taxila, Pakistan

DETAILED DESCRIPTION:
The main objective of this study is to assess the level of motivation towards physical activity and psychosocial outcomes (i.e., internalizing and externalizing behavioral symptoms, self-concept and academic achievement as assessed through recent grade) among young adolescents and to develop intervention to enhance motivation towards physical activity among young adolescents. Randomized Control Trial design will be used in this study to examine the impact of school-based intervention on motivation towards physical activity and psychosocial outcomes. After assessing their motivation toward physical activity and psychosocial outcomes intervention will given for 10 weeks, in which participants will be asked to participate in 10 minutes exercise activity on regular basis from Monday to Friday during school timings. Assessment will be done to find out that whether the school based intervention will be effective for them in motivation towards physical activity and reduction psychosocial outcomes (i.e., internalizing and externalizing behavioral symptoms, self-concept and academic achievement (as assessed through recent grade)) among adolescents or not. This results of this study will be used in promoting active lifestyle may help the adolescent to develop long-term positive healthy habits and targeting adolescents through encouraging physical activity in school or educational setting and social surrounding. To make decision about effective programs and policies to promote physical activity should be taken in account, by providing empirical support for public health messages that encourage participation in school spots as a mean to reduce the burden of poor mental health. Physical activity programming must align with the predictable developmental changes in adolescent exercise capacity and motor skills, which affect the activities in which they can successfully engage. These programs specifically designed to improve psychosocial outcomes, such as self-concept, social behavior and self-efficacy of adolescents as these are the most important determinants of participation in physical activities.

ELIGIBILITY:
Inclusion Criteria:

* Participants from grade 6th to 8th with in age range of 10-15 years.
* Participants who have lack of physical activity.
* Participants who provide consent to take part in the intervention.

Exclusion Criteria:

* Those participants who do not provide consent to take part in intervention will not be eligible take part in intervention.
* Participants who are having any physical disability or medical condition that compromises their mobility will not take part in intervention.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-12-10 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Motivation towards Physical Activity | 1 month
  the level of motivation towards physical activity will be assessed by the Participation Motivation Questionnaire.Participation Motivation Questionnaire is 3 point likert scale 1 for very important and 3 for not at all important.The Participation Motivation Questionnaire will revealed the factors of achievement/status, team atmosphere, fitness, energy release, skill development, friend- ship and fun as basic motives for involvement .
Level of Physical Activity | 1 month
  The Level of Physical Activity will be assessed through through using the physical activity questionnaire- adolescents (PAQ-A) is a self-administered, 7-day recall instrument , each scored on a 5-point scale. A score of 1 indicates low physical activity, whereas a score of 5 indicates high physical activity.
Psychosocial Outcomes | 1 month
  Psychosocial outcomes (i.e., internalizing and externalizing behavioral symptoms) will be assessed through Adolescents Behavioural Checklist is four point likert scale where o for Not at all and 3 for very much. Adolescents Behavioural Checklist consists of 48 items, 42 of which yield a total ABC score and six factor scores (Conduct Problems, Impulsivity/Hyperactivity, Poor Work Habits, Inattention, Emotional Liability, Social Problems).
Self Concept | 1 month
  Self-Concept will be assessed through using Self Concept Questionnaire .t consist of 48 items which provides 6 separate dimensions of self-concept (e.g physical, social, intellectual, moral, educational and temperamental) ,each item have 5 response.
Academic Achievement | 1 month
  Academic Achievement will be assess through recent academic achievement or performance in exams

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima Jinnah Women University Ethics Review Board, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No